CLINICAL TRIAL: NCT07003893
Title: Efficacy of Diaphragmatic Proprioceptive Neuromuscular Facilitation on Functional Capacity and Pulmonary Function in Heavy Twenties Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Zaytoonah University of Jordan (Other)
Responsible Party: Principal Investigator, Mohamed Saied Zidan, Assistant prof dr, Al-Zaytoonah University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB # 23/3/2024-2025
Record Dates: First submitted 2025-05-23; First posted 2025-06-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Smoking Dependence; Smoking Among Youth
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): perform exercises using aerobic exercises only
  Interventions: Other: Diaphragmatic Proprioceptive Neuromuscular Facilitation + Aerobic exercises
- Experimental group (Experimental): perform diaphragmatic proprioceptive neuromuscular facilitation and aerobic exercise
  Interventions: Other: Diaphragmatic Proprioceptive Neuromuscular Facilitation + Aerobic exercises

INTERVENTIONS:
Other: Diaphragmatic Proprioceptive Neuromuscular Facilitation + Aerobic exercises — Control group will perform aerobic exercises only Experimental group will perform diaphragmatic proprioceptive neuromuscular facilitation in addition to aerobic exercises

SUMMARY:
Although research on the health risks of e-cigarettes is still limited, there is increasing evidence of debilitating lung disease and general immune dysfunction from e-cigarettes, leading to various infections. Moreover, there are concerns that e-cigarettes can cause general impairment in life functions and more importantly lung function .Although exercise can help quit smoking and reduce relapses .However, exercise has many other fitness benefits when done regularly for the general population, as well as for smokers. Exercise has been shown to help with smoking cessation, which has been an important factor preventing many smokers, especially younger people, from quitting. Breathing exercises, especially diaphragm exercises improves lung function, lifestyle and health risk factors and thus the risk of developing many chronic diseases. Both aerobic interventions and exercise can reduce the incidence of many of the prevalent cancers initiated by smoking, such as lung cancer. This is important because lung cancer is the most common type of cancer worldwide, and cigarette smoking is responsible for up to 90% of lung cancer cases worldwide.

DETAILED DESCRIPTION:
According to predictions by the World Health Organization, the number of smokers who will die from cigarette related diseases will surpass the number of people dying from AIDS, traffic accidents, suicide, and murder combined by 2020. Due to the presence of various harmful substances in cigarettes, smoking can cause many diseases. Nicotine which is one of the major constituents of cigarettes causes arteriosclerosis, coronary artery disease, chronic obstructive pulmonary disease (COPD), and other problems that result not only in low cardiopulmonary function but also in relatively diminished daily living ability and endurance in smokers compared with that in non-smokers. Moreover, it is common knowledge that smoking is very highly correlated with occurrence of respiratory diseases. Diaphragmatic breathing is a good technique for respiration and relaxation of the lungs because it enables sufficient exchange of oxygen and carbon dioxide. Diaphragmatic breathing is reported to be effective in improvement of ventilation efficiency, dyspnea, and activity ability; reduction of metabolic acidosis; alleviation of back pain; spine correction; abdominal strengthening; and improvement of body composition and flexibility. In our current social climate, the number of male smokers in their twenties is rapidly increasing and this trend is becoming a social problem. Our study attempts to verify the effects of diaphragmatic proprioceptive neuromuscular facilitation on functional capacity and pulmonary functions in in heavy twenties smokers.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20-29 years.

  * Subjects who have been smoking for 1 to 3 years.
  * Subjects who not receiving medical treatment for respiratory diseases.
  * Subjects who have clean family medical history.

Exclusion Criteria:

* Subjects who smoke cigars other than filtered cigarettes or tobacco pipes.

  * Subjects with respiratory proplems.
  * Participation in another clinical trial within the last 30 days.
  * Endocrine and metabolic disorders (eg, hypothyroidism, hypercalcemia, diabetes mellitus, diabetes insipidus).
  * Neurologic and psychiatric disorders (who can not understand the research project ).

Ages: 20 Years to 29 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2025-07-05 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-02 (Actual)

PRIMARY OUTCOMES:
FEV1/FVC ( % ) | pre and post 4 weeks
  The ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lungs. That can reflect pulmonary function , using portable spirometer ( SP 80B,China)
FEV1 ( liters ) | Pre and post 4 weeks
  Forced expiratory volume in 1 second that can reflect pulmonary function , using portable spirometer ( SP 80B,China)
PEF ( liters / minute ) | pre and post 4 weeks
  Peak expiratory flow (PEF), a key indicator of lung function,using portable spirometer ( SP 80B,China)
FVC ( liters ) | Pre and post 4 weeks
  Forced vital capacity (FVC) is the total amount of air exhaled during the FEV test. Forced expiratory volume and forced vital capacity are lung function tests , using portable spirometer ( SP 80B , China )
Chest expansion ( centimeter ) | Pre and post 4 weeks
  A simple, noninvasive pulmonary function test used to assess chest wall mobility and, to a lesser extent, lung function , using tape measurement.

SECONDARY OUTCOMES:
Functional capacity | Pre and post 4 weeks
  By using 6MWDT

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Saied Zidan, Cairo, Egypt